CLINICAL TRIAL: NCT03847389
Title: Open-Label Study of the Pharmacokinetics and Safety Including HPA Axis Suppression Potential of Clobetasol Topical Oil in Pediatric Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: Clobetasol Topical Oil for Children With Moderate to Severe Atopic Dermatitis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Difficulty in enrollment and COVID-19 pandemic.
Sponsor: Hill Dermaceuticals, Inc. (Industry)
Collaborators: Synteract, Inc. (Industry); Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP0418 SS-P2 051
Record Dates: First submitted 2019-01-23; First posted 2019-02-20 (Actual); Results first posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Clobetasol; Oils

STUDY DESIGN:
Intervention Model Description: open-label, maximal use, in 3 successive age cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- clobetasol propionate topical oil (Other): clobetasol propionate 0.05% topical oil applied as thin film twice daily for 2 weeks
  Interventions: Drug: Clobetasol propionate 0.05% Topical Oil

INTERVENTIONS:
Drug: Clobetasol propionate 0.05% Topical Oil — thin film application of the oil twice daily
  Other Names: clobetasol propionate topical solution

SUMMARY:
Open-Label Study designed to evaluate the HPA axis suppression potential of Clobetasol Topical Oil and pharmacokinetic safety / systemic exposure to clobetasol when Clobetasol Topical Oil is applied to pediatric subjects with moderate to severe atopic dermatitis (AD) under maximal use conditions.

The study duration for each subject will be up to 54 days (up to 38 days for Screening assessments, followed by up to 16 days of treatment and follow-up). Additional time will be required for subjects requiring additional hypothalamic-pituitary-adrenal [HPA] axis function testing due to an abnormal result at End of Treatment.

DETAILED DESCRIPTION:
This study is a multicenter, open-label study designed to evaluate the HPA axis suppression potential and systemic exposure to clobetasol, when administered as Clobetasol Topical Oil in pediatric subjects, under conditions consistent with anticipated clinical use and under conditions designed to maximize the potential for drug absorption in subjects with moderate to severe AD. The study will consist of three successively younger pediatric cohorts, as safety data allow:

* Cohort 1: ≥12 to <18 years;
* Cohort 2: ≥6 to <12 years; and
* Cohort 3: ≥2 to <6 years. Enrollment into each successively younger pediatric cohort will proceed only after the preceding cohort has been completed and safety and exploratory data (including adverse events [AEs], tolerability assessments, clinical laboratory results, and the percentage of subjects with HPA axis suppression) have been reviewed and agreed to be acceptable for progression to the next cohort. Enrollment into Cohorts 2 and 3 will proceed only if the percentage of subjects with HPA axis suppression in Cohorts 1 and 2, respectively, is ≤40%. HPA axis suppression is defined as a cortisol concentration ≤18 µg/100 mL at approximately 30 minutes after stimulation with cosyntropin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects in good general health confirmed by medical history.
* Subjects with a clinical diagnosis of AD (according to the criteria of Hanifin and Rajka) of moderate to severe intensity (ISGA score of 3 or 4) involving ≥25% to ≤50% of total BSA located within treatable areas (Cohort 1), or ≥35% to ≤50% of total BSA located within treatable areas (Cohorts 2 and 3), with treatable areas including all but the face, axillae, groin, and scalp.
* Subjects with a normally functioning HPA axis, defined as a prestimulation serum cortisol level >5 µg/100 mL, and a response to cosyntropin stimulation to >18 µg/100 mL (after approximately 30 minutes); both blood draws for this test should be performed in the morning, if possible
* Female subjects of childbearing potential must have a negative urine pregnancy test, must not be breastfeeding, and must agree to use an acceptable form of birth control for the duration of the study. Female subjects of childbearing potential are defined as all female subjects who have reached menarche and are not two years postmenopausal or who have reached menarche and have not had a hysterectomy, bilateral tubal ligation, and/or complete bilateral oophorectomy

Exclusion Criteria:

* Subjects who do not have a normally functioning HPA axis (as defined in the inclusion criteria).
* Subjects with an abnormal sleep schedule or who work at night.
* Subjects who have used topical dermal corticosteroids or topical immunomodulators (e.g., tacrolimus or pimecrolimus) within 3 weeks before Day 1, and subjects who are using any systemic medication known to affect cortisol levels or HPA axis integrity, systemic corticosteroids, an acute systemic course of corticosteroids, and/or any biological medication within 30 days before Day 1.
* Subjects with concomitant medical or dermatologic disorders (neurodermatitis, skin atrophy, striae, telangiectasia, etc.) that may interfere with study objectives and/or evaluations.
* Subjects with active skin infection.
* Subjects with any known significant endocrinological disorder that may require prohibited treatment, any known underlying disease that the investigator deems uncontrolled and poses a safety risk for the subject while participating in the study, known sensitivity to any ingredient of the study preparation, or a history of adverse responses to topical or systemic steroid therapy.
* Subjects who are pregnant or nursing.
* Subjects who have used bleach baths, phototherapy, and/or tanning beds, and/or who have had excessive sun exposure within 1 week before Day 1 and/or are planning to use any of these during the study.
* Subjects who have participated in a clinical drug or device research study and/or used any investigational treatment within the last 30 days before Day

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-05-02 (Actual); Study Completion 2020-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosario G Ramirez, MD, Study Director — Hill Dermaceuticals, Inc.
Locations (6):
- United States (6):
  - International Clinical Research - US, LLC, Sanford, Florida
  - AeroAllergy Research Laboratories of Savannah, Inc, Savannah, Georgia
  - Paddington Testing Co., Inc., Philadelphia, Pennsylvania
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Progressive Clinical Research, San Antonio, Texas
  - Clinical Research Partners, LLC, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment into each successively younger pediatric cohort was to proceed only after the preceding cohort had been completed, and safety and exploratory data reviewed and agreed to be acceptable for progression to the next cohort. Enrollment into Cohorts 2 and 3 proceeded only if the subjects with HPA axis suppression in Cohorts 1 and 2, respectively, was ≤40%.
Groups:
- Clobetasol Propionate Topical Oil in Cohort 1: Cohort 1: ≥12 to <18 years;
  Enrollment into each successively younger pediatric cohort was to have proceeded only after the preceding cohort had been completed and safety and exploratory data (including adverse events [AEs], tolerability assessments, clinical laboratory results, and the percentage of subjects with HPA axis suppression) had been reviewed and agreed to be acceptable for progression to the next cohort. Enrollment into Cohorts 2 and 3 were to have proceeded only if the percentage of subjects with HPA axis suppression in Cohorts 1 and 2, respectively, was ≤40%. HPA axis suppression was defined as a cortisol concentration ≤18 µg/100 mL at approximately 30 minutes after stimulation with cosyntropin.
- Clobetasol Propionate Topical Oil in Cohort 2: Cohort 2: ≥6 to <12 years;
  Enrollment into each successively younger pediatric cohort was to have proceeded only after the preceding cohort had been completed and safety and exploratory data (including adverse events [AEs], tolerability assessments, clinical laboratory results, and the percentage of subjects with HPA axis suppression) had been reviewed and agreed to be acceptable for progression to the next cohort. Enrollment into Cohorts 2 and 3 were to have proceeded only if the percentage of subjects with HPA axis suppression in Cohorts 1 and 2, respectively, was ≤40%. HPA axis suppression was defined as a cortisol concentration ≤18 µg/100 mL at approximately 30 minutes after stimulation with cosyntropin.
- Clobetasol Propionate Topical Oil in Cohort 3: Cohort 3: ≥2 to <6 years
  Enrollment into each successively younger pediatric cohort was to have proceeded only after the preceding cohort had been completed and safety and exploratory data (including adverse events [AEs], tolerability assessments, clinical laboratory results, and the percentage of subjects with HPA axis suppression) had been reviewed and agreed to be acceptable for progression to the next cohort. Enrollment into Cohorts 2 and 3 were to have proceeded only if the percentage of subjects with HPA axis suppression in Cohorts 1 and 2, respectively, was ≤40%. HPA axis suppression was defined as a cortisol concentration ≤18 µg/100 mL at approximately 30 minutes after stimulation with cosyntropin.
Period: Overall Study
Arm/Group | Clobetasol Propionate Topical Oil in Cohort 1 | Clobetasol Propionate Topical Oil in Cohort 2 | Clobetasol Propionate Topical Oil in Cohort 3
Started | 8 | 0 (Start of Cohort 2 can only happen if less than or equal to 40% of subjects in Cohort 1 had HPA axis suppression.) | 0 (Start of Cohort 3 can only happen if less than or equal to 40% of subjects in Cohort 2 had HPA axis suppression.)
Completed | 8 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated prior to enrolling participants in cohort 2 or cohort 3.
Groups:
- Clobetasol Propionate Topical Oil in Cohort 1: Cohort 1: ≥12 to <18 years;
  At the Baseline/Start of Treatment for Cohort 1, subjects underwent assessments of their AD, baseline (pretreatment) assessments of tolerability criteria, a review of eligibility criteria, a urine pregnancy test and baseline (pretreatment) assessments of AEs. For subjects who remained eligible for the study, the investigator designated the areas to be treated with study drug, and subjects and/or their caregivers applied the first dose of study drug at the site. AEs and tolerability were assessed.
- Clobetasol Propionate Topical Oil in Cohort 2: Cohort 2: ≥6 to <12 years;
  Enrollment from Cohort 1 into Cohort 2 will proceed only after cohort 1 had been completed and safety and exploratory data (including adverse events [AEs], tolerability assessments, clinical laboratory results, and the percentage of subjects with HPA axis suppression) had been reviewed and agreed to be acceptable, and only if the percentage of subjects with HPA axis suppression in Cohort 1 was ≤40%. HPA axis suppression was defined as a cortisol concentration ≤18 µg/100 mL at approximately 30 minutes after stimulation with cosyntropin.
- Clobetasol Propionate Topical Oil in Cohort 3: Cohort 3: ≥2 to <6 years
  Enrollment from Cohort 2 into Cohort 3 will proceed only after cohort 2 had been completed and safety and exploratory data (including adverse events [AEs], tolerability assessments, clinical laboratory results, and the percentage of subjects with HPA axis suppression) had been reviewed and agreed to be acceptable, and only if the percentage of subjects with HPA axis suppression in Cohort 1 was ≤40%. HPA axis suppression was defined as a cortisol concentration ≤18 µg/100 mL at approximately 30 minutes after stimulation with cosyntropin.
- Total: Total of all reporting groups
Arm/Group | Clobetasol Propionate Topical Oil in Cohort 1 | Clobetasol Propionate Topical Oil in Cohort 2 | Clobetasol Propionate Topical Oil in Cohort 3 | Total
Number analyzed (Participants) | 8 | 0 | 0 | 8
Age, Continuous [Median (Full Range); unit: years] | 17 [12 to 18] |  |  | 17 [12 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 |  |  | 6
  Male | 2 |  |  | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 |  |  | 4
  Not Hispanic or Latino | 4 |  |  | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 |  |  | 8
prestimulation serum cortisol level >5 µg/100 mL, [Count of Participants; unit: Participants] | 8 |  |  | 8
post-stimulation cortisol level >18 µg/100 mL [Count of Participants; unit: Participants] | 8 |  |  | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With HPA Axis Suppression - Serum Cortisol Concentration (Cortrosyn Stimulation Test)
Description: 30-minute Post-stimulation cortisol level ≤18 µg/100 mL at Day 0 means subject is not enrolled; 30-minute Post-stimulation cortisol level ≤18 µg/100 mL at end of treatment (Day 15) means subject had suppression.
Time Frame: day 0 and day 15.
Population: Subjects met all eligibility criteria and were enrolled. Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Clobetasol Propionate Topical Oil in Cohort 1 | Clobetasol Propionate Topical Oil in Cohort 2 | Clobetasol Propionate Topical Oil in Cohort 3
Number analyzed (Participants) | 8 | 0 | 0
Participants
  Subjects with post-stimulation cortisol level ≤18 µg/100 mL at Day 0 (before treatment) | 0 | 0 | 0
  Subjects with post-stimulation cortisol level ≤18 µg/100 mL at any time during treatment | 3 | 0 | 0
  Subjects with post-stimulation cortisol level greater than18 µg/100 mL at end of treatment (Day 15) | 5 |  |

2. Primary Outcome: Adverse Events, Including Treatment Emergent Adverse Events (TEAEs)
Description: number of events and percentage of subjects with AEs including TEAEs
Time Frame: Days 0, 1, 8 and 15
Population: All subjects who met eligibility criteria for enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Clobetasol Propionate Topical Oil in Cohort 1 | Clobetasol Propionate Topical Oil in Cohort 2 | Clobetasol Propionate Topical Oil in Cohort 3
Number analyzed (Participants) | 8 | 0 | 0
Participants
  Subjects without AEs, including treatment emergent adverse events | 8 | 0 | 0
  Subjects with AEs | 0 | 0 | 0

3. Other Pre Specified Outcome: ISGA Category
Description: ISGA results will be summarized at each visit as:
  1. number and percentage of subjects in each ISGA category
  2. number and percentage of subjects with an ISGA score of either 0 or 1 (clear or almost clear)
  3. number and percentage of subjects with an ISGA improvement of at least 2 grades from Baseline to each post-baseline evaluation
  4. number and percentage of subjects with an ISGA score of either 0 or 1 (clear or almost clear) and an improvement of at least 2 grades from Baseline to each post-Baseline evaluation
Time Frame: Days 0, 1, 8 and 15 Efficacy assessment, including ISGA, was not performed due to premature termination of the study.
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Assessment of Burning/Stinging, Skin Atrophy, Striae, Folliculitis, and Telangiectasias (Tolerability Parameters).
Description: The subject will rate the sensation of burning/stinging within the past 24 hours as none (0), mild (1), moderate (2) or severe (3), and the Investigator will assess skin atrophy, striae, folliculitis, and telangiectasias, as absent (0) or present (1).
Time Frame: Days 1, 8 and 15
Population: All subjects that met eligibility criteria for enrollment. Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Clobetasol Propionate Topical Oil in Cohort 1 | Clobetasol Propionate Topical Oil in Cohort 2 | Clobetasol Propionate Topical Oil in Cohort 3
Number analyzed (Participants) | 8 | 0 | 0
Participants
  No AEs | 8 |  |
  With AEs | 0 |  |

ADVERSE EVENTS:
Time Frame: AEs were collected at start of study to termination of the study, approximately 6 months.
Description: All adverse events (AEs) which started after the start of study drug or which increased from baseline in severity were considered treatment emergent AEs (TEAEs).
Arm/Group | Clobetasol Propionate Topical Oil in Cohort 1 | Clobetasol Propionate Topical Oil in Cohort 2 | Clobetasol Propionate Topical Oil in Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/8 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated early due to the COVID pandemic with very low subject enrollment. Due to the small number of subjects that completed when the study was prematurely terminated, pharmacokinetic, exploratory, sensitivity, as well as some safety analyses was not completed under the SAP.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT03847389/Prot_002.pdf
  • Statistical Analysis Plan (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT03847389/SAP_001.pdf